CLINICAL TRIAL: NCT06160583
Title: General Anesthesia in Obstetric Patients for Cesarean Section, Maternal and Perinatal Outcomes
Brief Title: General Anesthesia for Cesarean Section, Maternal and Perinatal Outcomes
Status: Completed | Type: Observational
Sponsor: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Diego Francisco Gonzalez Pena, Anestesiologist, Hospital Civil de Guadalajara
Other Study IDs: 257/23
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Anesthesia; Perinatal Morbidity; Maternal-Fetal Relations
Keywords: General anesthesia; Materno; Perinatal; Outcomes; Cesarean

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the maternal and perinatal outcomes that occur in obstetric patients undergoing cesarean section surgery under general anesthesia at the Fray Antonio Alcalde Civil Hospital of Guadalajara.

DETAILED DESCRIPTION:
Pregnant patients who required surgical management to resolve the pregnancy via the abdominal route will be identified from the anesthesiology logs and evaluation sheets of the obstetric patient. During the period from January 2019 to December 2023.

The data will be collected in a database made up of Excel software. Maternal data collected:Of the total cesarean surgery procedures, the following are collected: hospital record, the anesthetic technique administered and the date of the surgical intervention.

Patients who underwent surgery under general anesthesia technique will be identified and their demographic data will be recorded (name, age, hospital record, weight, height, BMI, obstetric data, number of pregnancies, births, cesarean sections, abortions, weeks of gestation) diagnosis. , type of intervention, procedure performed The characteristics of the anesthetic technique, the drugs used for anesthetic induction, will also be recorded.

Complications associated with the anesthetic technique will be recorded, such as: intraoperative awakening, failed tracheal intubation and pulmonary aspiration.

The status of the patient's discharge from the operating room, extubated or intubated, will be recorded.

Fetal data collected: Prenatal fetal diagnosis will be obtained, as well as its classification by ultrasound measurement of estimated weight and weeks of gestation assigned to weight appropriate for gestational age, small for gestational age or large for gestational age.

From the results of the newborn, the condition at birth, weight, height, gestational age, as well as the size at birth assigned in: adequate weight, low or high, are recorded.

The Apgar score will be obtained at one minute and at 5 minutes. The condition of the newborn after immediate care will be recorded if he or she remains in rooming-in or is discharged to surveillance, intermediate or intensive therapy.

Data that is not found in the obstetric patient's evaluation sheets will be corroborated in anesthesiology, nursing, neonatology logs and electronic records. Once the database is obtained, the statistical analysis will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Obstetric patients who require surgical intervention to resolve the pregnancy, under general anesthesia

Exclusion Criteria:

* Obstetric patients who enter the hospital intubated.

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Obstetric patients
Study Population: Obstetric patients who require cesarean section surgery at the Fray Antonio Alcalde Civil Hospital of Guadalajara
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2023-11-12 (Actual); Primary Completion 2023-11-12 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Frequency general anesthesia | 5 years
  Obtain the frequency of obstetric patients undergoing cesarean section surgery under general anesthesia
Maternal and fetal diagnosis | 5 years
  Specify the diagnoses for which general anesthesia is carried out
Classification physical status | 5 years
  Know the physical status of patients undergoing cesarean surgery
General anesthesia complications | 5 years
  Identify complications of the anesthetic technique
Maternal condition at the end of surgery | 5 years
  List the maternal discharge condition at the end of surgery (intubated/extubated)
Anesthetic induction | 5 years
  Describe the medications used for anesthetic induction
Prenatal classification by weight and gestational age | 5 years
  Document prenatal classification of the fetus by weight and gestational age assigned by ultrasound
Apgar Score | 5 years
  Record the newborn's Apgar score Apgar scale It evaluates a score from 0 to 10, the higher the score, the better the baby's progress. a score greater than 7 is considered normal
Size at birth | 5 years
  Document birth size classification assigned by neonatology
Condition of the newborn | 5 years
  List the condition of the newborn after his or her initial evaluation (rooming-in/neonatal therapy)

CONTACTS AND LOCATIONS:
Overall Officials: Diego Francisco Gonzalez Peña, MD, Principal Investigator — Hospital Civil de Guadalajara; María de los Angeles Campechano Ascencio, MSc, Study Director — Hospital Civil de Guadalajara; Jorge Bravo Rubio, PhD, Study Chair — Hospital Civil de Guadalajara; Ofelia Margarita Ascencio Aceves, MD, Study Chair — Hospital Civil de Guadalajara
Locations (1):
- Maria de Los Angeles Campechano Ascencio, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No
The records collected will be used exclusively for the results of this protocol

REFERENCES:
- [Result] Mhyre JM, Sultan P. General Anesthesia for Cesarean Delivery: Occasionally Essential but Best Avoided. Anesthesiology. 2019 Jun;130(6):864-866. doi: 10.1097/ALN.0000000000002708. No abstract available. PMID 30985305
- [Result] Ikeda T, Kato A, Bougaki M, Araki Y, Ohata T, Kawashima S, Imai Y, Ninagawa J, Oba K, Chang K, Uchida K, Yamada Y. A retrospective review of 10-year trends in general anesthesia for cesarean delivery at a university hospital: the impact of a newly launched team on obstetric anesthesia practice. BMC Health Serv Res. 2020 May 13;20(1):421. doi: 10.1186/s12913-020-05314-2. PMID 32404093
- [Result] Kodali BS, Chandrasekhar S, Bulich LN, Topulos GP, Datta S. Airway changes during labor and delivery. Anesthesiology. 2008 Mar;108(3):357-62. doi: 10.1097/ALN.0b013e31816452d3. PMID 18292672
- [Result] Robbins LS, Blanchard CT, Biasini FJ, Powell MF, Casey BM, Tita AT, Harper LM. General anesthesia for cesarean delivery and childhood neurodevelopmental and perinatal outcomes: a secondary analysis of a randomized controlled trial. Int J Obstet Anesth. 2021 Feb;45:34-40. doi: 10.1016/j.ijoa.2020.08.007. Epub 2020 Aug 25. PMID 33121885
- [Result] Bowring J, Fraser N, Vause S, Heazell AE. Is regional anaesthesia better than general anaesthesia for caesarean section? J Obstet Gynaecol. 2006 Jul;26(5):433-4. doi: 10.1080/01443610600720345. PMID 16846870
- [Result] Lumbiganon P, Moe H, Kamsa-Ard S, Rattanakanokchai S, Laopaiboon M, Kietpeerakool C, Jampathong N, Somjit M, Cecatti JG, Vogel JP, Betran AP, Mittal S, Torloni MR. Outcomes associated with anaesthetic techniques for caesarean section in low- and middle-income countries: a secondary analysis of WHO surveys. Sci Rep. 2020 Jun 23;10(1):10176. doi: 10.1038/s41598-020-66897-8. PMID 32576845
- [Result] Metogo JAM, Nana TN, Ngongheh BA, Nyuydzefon EB, Adjahoung CA, Tochie JN, Minkande JZ. General versus regional anaesthesia for caesarean section indicated for acute foetal distress: a retrospective cohort study. BMC Anesthesiol. 2021 Mar 4;21(1):68. doi: 10.1186/s12871-021-01289-7. PMID 33663391
- [Result] Swanson K, Liang L, Grobman WA, Higgins N, Roy A, Son M. Duration of Exposure to General Endotracheal Anesthesia during Cesarean Deliveries at Term and Perinatal Complications. Am J Perinatol. 2022 Feb;39(3):232-237. doi: 10.1055/s-0041-1739355. Epub 2021 Nov 29. PMID 34844279
- [Result] Ozden MGN, Koruk S, Collak Z, Panik N. Comparison of the effects of general and spinal anesthesia for cesarean delivery on maternal and fetal outcomes: A retrospective analysis of data. North Clin Istanb. 2023 Sep 11;10(5):575-582. doi: 10.14744/nci.2023.25593. eCollection 2023. PMID 37829746
- [Result] Devroe S, Van de Velde M, Rex S. General anesthesia for caesarean section. Curr Opin Anaesthesiol. 2015 Jun;28(3):240-6. doi: 10.1097/ACO.0000000000000185. PMID 25827280
- [Result] Neef V, Wenk M, Kranke P. [Obstetric Anesthesia]. Anasthesiol Intensivmed Notfallmed Schmerzther. 2023 Oct;58(10):570-582. doi: 10.1055/a-2043-4329. Epub 2023 Oct 13. German. PMID 37832560
- [Result] Munro A, Sjaus A. General anesthesia for Cesarean delivery: can interinstitutional variation in practice offer deeper insights into our choice of anesthetic modality? Can J Anaesth. 2024 Feb;71(2):169-174. doi: 10.1007/s12630-023-02634-9. Epub 2023 Nov 6. No abstract available. PMID 37932651
- [Result] Mushambi MC, Kinsella SM, Popat M, Swales H, Ramaswamy KK, Winton AL, Quinn AC; Obstetric Anaesthetists' Association; Difficult Airway Society. Obstetric Anaesthetists' Association and Difficult Airway Society guidelines for the management of difficult and failed tracheal intubation in obstetrics. Anaesthesia. 2015 Nov;70(11):1286-306. doi: 10.1111/anae.13260. PMID 26449292
- [Result] Munnur U, de Boisblanc B, Suresh MS. Airway problems in pregnancy. Crit Care Med. 2005 Oct;33(10 Suppl):S259-68. doi: 10.1097/01.ccm.0000183502.45419.c9. PMID 16215346
- [Result] Jain K, Gupta N, Yadav M, Thulkar S, Bhatnagar S. Radiological evaluation of airway - What an anaesthesiologist needs to know! Indian J Anaesth. 2019 Apr;63(4):257-264. doi: 10.4103/ija.IJA_488_18. PMID 31000888
- [Result] Wise RA, Polito AJ, Krishnan V. Respiratory physiologic changes in pregnancy. Immunol Allergy Clin North Am. 2006 Feb;26(1):1-12. doi: 10.1016/j.iac.2005.10.004. PMID 16443140
- [Result] Dallmann A, Ince I, Meyer M, Willmann S, Eissing T, Hempel G. Gestation-Specific Changes in the Anatomy and Physiology of Healthy Pregnant Women: An Extended Repository of Model Parameters for Physiologically Based Pharmacokinetic Modeling in Pregnancy. Clin Pharmacokinet. 2017 Nov;56(11):1303-1330. doi: 10.1007/s40262-017-0539-z. PMID 28401479
- [Result] Sanghavi M, Rutherford JD. Cardiovascular physiology of pregnancy. Circulation. 2014 Sep 16;130(12):1003-8. doi: 10.1161/CIRCULATIONAHA.114.009029. No abstract available. PMID 25223771
- [Result] Sung S, Mikes BA, Martingano DJ, Mahdy H. Cesarean Delivery. 2024 Dec 7. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK546707/ PMID 31536313
- [Result] Cobb BT, Lane-Fall MB, Month RC, Onuoha OC, Srinivas SK, Neuman MD. Anesthesiologist Specialization and Use of General Anesthesia for Cesarean Delivery. Anesthesiology. 2019 Feb;130(2):237-246. doi: 10.1097/ALN.0000000000002534. PMID 30601216
- [Result] Dahlke JD, Mendez-Figueroa H, Rouse DJ, Berghella V, Baxter JK, Chauhan SP. Evidence-based surgery for cesarean delivery: an updated systematic review. Am J Obstet Gynecol. 2013 Oct;209(4):294-306. doi: 10.1016/j.ajog.2013.02.043. Epub 2013 Mar 1. PMID 23467047
- [Result] Betran AP, Ye J, Moller AB, Zhang J, Gulmezoglu AM, Torloni MR. The Increasing Trend in Caesarean Section Rates: Global, Regional and National Estimates: 1990-2014. PLoS One. 2016 Feb 5;11(2):e0148343. doi: 10.1371/journal.pone.0148343. eCollection 2016. PMID 26849801
- [Result] Al Rifai RH. Trend of caesarean deliveries in Egypt and its associated factors: evidence from national surveys, 2005-2014. BMC Pregnancy Childbirth. 2017 Dec 13;17(1):417. doi: 10.1186/s12884-017-1591-2. PMID 29237410
- [Result] Butwick AJ, Palanisamy A. Mode of anaesthesia for Caesarean delivery and maternal morbidity: can we overcome confounding by indication? Br J Anaesth. 2018 Apr;120(4):621-623. doi: 10.1016/j.bja.2018.01.002. Epub 2018 Feb 14. No abstract available. PMID 29576102
- [Result] Elnakib S, Abdel-Tawab N, Orbay D, Hassanein N. Medical and non-medical reasons for cesarean section delivery in Egypt: a hospital-based retrospective study. BMC Pregnancy Childbirth. 2019 Nov 8;19(1):411. doi: 10.1186/s12884-019-2558-2. PMID 31703638
- [Result] Schatz M, Dombrowski MP. Clinical practice. Asthma in pregnancy. N Engl J Med. 2009 Apr 30;360(18):1862-9. doi: 10.1056/NEJMcp0809942. No abstract available. PMID 19403904
- [Result] Bonhomme V, Staquet C, Montupil J, Defresne A, Kirsch M, Martial C, Vanhaudenhuyse A, Chatelle C, Larroque SK, Raimondo F, Demertzi A, Bodart O, Laureys S, Gosseries O. General Anesthesia: A Probe to Explore Consciousness. Front Syst Neurosci. 2019 Aug 14;13:36. doi: 10.3389/fnsys.2019.00036. eCollection 2019. PMID 31474839
- [Result] Siddik-Sayyid S, Zbeidy R. Practice guidelines for obstetric anesthesia--a summary. Middle East J Anaesthesiol. 2008 Oct;19(6):1291-303. No abstract available. PMID 18942244
- [Result] Franks NP. General anaesthesia: from molecular targets to neuronal pathways of sleep and arousal. Nat Rev Neurosci. 2008 May;9(5):370-86. doi: 10.1038/nrn2372. PMID 18425091
- [Result] McGuire B, Lucas DN. Planning the obstetric airway. Anaesthesia. 2020 Jul;75(7):852-855. doi: 10.1111/anae.14987. Epub 2020 Mar 6. No abstract available. PMID 32144754
- [Result] Juang J, Gabriel RA, Dutton RP, Palanisamy A, Urman RD. Choice of Anesthesia for Cesarean Delivery: An Analysis of the National Anesthesia Clinical Outcomes Registry. Anesth Analg. 2017 Jun;124(6):1914-1917. doi: 10.1213/ANE.0000000000001677. PMID 28098588
- [Result] Ring L, Landau R, Delgado C. The Current Role of General Anesthesia for Cesarean Delivery. Curr Anesthesiol Rep. 2021;11(1):18-27. doi: 10.1007/s40140-021-00437-6. Epub 2021 Feb 24. PMID 33642943
- [Result] Husarova V, McCaul CL. Incidence of general anaesthesia for caesarean section in parturients from different geographic regions: 7-year retrospective study in a single European university centre. Eur J Anaesthesiol. 2016 Jun;33(6):466-8. doi: 10.1097/EJA.0000000000000396. No abstract available. PMID 26840830
- [Result] Al-Husban N, Elmuhtaseb MS, Al-Husban H, Nabhan M, Abuhalaweh H, Alkhatib YM, Yousef M, Aloran B, Elyyan Y, Alghazo A. Anesthesia for Cesarean Section: Retrospective Comparative Study. Int J Womens Health. 2021 Feb 2;13:141-152. doi: 10.2147/IJWH.S292434. eCollection 2021. PMID 33564269
- [Result] Detsky ME, Jivraj N, Adhikari NK, Friedrich JO, Pinto R, Simel DL, Wijeysundera DN, Scales DC. Will This Patient Be Difficult to Intubate?: The Rational Clinical Examination Systematic Review. JAMA. 2019 Feb 5;321(5):493-503. doi: 10.1001/jama.2018.21413. PMID 30721300
- [Result] Preston R, Jee R. Obstetric airway management. Int Anesthesiol Clin. 2014 Spring;52(2):1-28. doi: 10.1097/AIA.0000000000000014. No abstract available. PMID 24667446
- [Result] Sumikura H, Niwa H, Sato M, Nakamoto T, Asai T, Hagihira S. Rethinking general anesthesia for cesarean section. J Anesth. 2016 Apr;30(2):268-73. doi: 10.1007/s00540-015-2099-4. Epub 2015 Nov 19. PMID 26585767
- [Result] Sajayan A, Wicker J, Ungureanu N, Mendonca C, Kimani PK. Current practice of rapid sequence induction of anaesthesia in the UK - a national survey. Br J Anaesth. 2016 Sep;117 Suppl 1:i69-i74. doi: 10.1093/bja/aew017. Epub 2016 Feb 24. PMID 26917599
- [Result] McNarry AF, Patel A. The evolution of airway management - new concepts and conflicts with traditional practice. Br J Anaesth. 2017 Dec 1;119(suppl_1):i154-i166. doi: 10.1093/bja/aex385. PMID 29161401
- [Result] Delgado C, Ring L, Mushambi MC. General anaesthesia in obstetrics. BJA Educ. 2020 Jun;20(6):201-207. doi: 10.1016/j.bjae.2020.03.003. Epub 2020 Apr 21. No abstract available. PMID 33456951
- [Result] Maronge L, Bogod D. Complications in obstetric anaesthesia. Anaesthesia. 2018 Jan;73 Suppl 1:61-66. doi: 10.1111/anae.14141. PMID 29313912
- [Result] Guglielminotti J, Landau R, Li G. Adverse Events and Factors Associated with Potentially Avoidable Use of General Anesthesia in Cesarean Deliveries. Anesthesiology. 2019 Jun;130(6):912-922. doi: 10.1097/ALN.0000000000002629. PMID 30789362
- [Result] D'Angelo R, Smiley RM, Riley ET, Segal S. Serious complications related to obstetric anesthesia: the serious complication repository project of the Society for Obstetric Anesthesia and Perinatology. Anesthesiology. 2014 Jun;120(6):1505-12. doi: 10.1097/ALN.0000000000000253. PMID 24845921
- [Result] Aydas AD, Basaranoglu G, Ozdemir H, Dooply SL, Muhammedoglu N, Kucuk S, Saidoglu L. Airway changes in pregnant women before and after delivery. Ir J Med Sci. 2015 Jun;184(2):431-3. doi: 10.1007/s11845-014-1138-8. Epub 2014 May 24. PMID 24859287
- [Result] Committee Opinion No. 644: The Apgar Score. Obstet Gynecol. 2015 Oct;126(4):e52-e55. doi: 10.1097/AOG.0000000000001108. PMID 26393460
- [Result] Hassanin AS, El-Shahawy HF, Hussain SH, Bahaa Eldin AM, Elhawary MM, Elbakery M, Elsafty MSE. Impact of interval between induction of spinal anesthesia to delivery on umbilical arterial cord ph of neonates delivered by elective cesarean section. BMC Pregnancy Childbirth. 2022 Mar 17;22(1):216. doi: 10.1186/s12884-022-04536-y. PMID 35300620
- [Result] Garcia-Alix Perez A. [Non-reassuring fetal status, perinatal asphyxia and neonatal encephalopathy]. An Pediatr (Barc). 2005 Jul;63(1):1-4. doi: 10.1157/13076760. No abstract available. Spanish. PMID 15989864
- [Result] Salomon LJ, Alfirevic Z, Da Silva Costa F, Deter RL, Figueras F, Ghi T, Glanc P, Khalil A, Lee W, Napolitano R, Papageorghiou A, Sotiriadis A, Stirnemann J, Toi A, Yeo G. ISUOG Practice Guidelines: ultrasound assessment of fetal biometry and growth. Ultrasound Obstet Gynecol. 2019 Jun;53(6):715-723. doi: 10.1002/uog.20272. PMID 31169958
- [Result] Hollowell J, Pillas D, Rowe R, Linsell L, Knight M, Brocklehurst P. The impact of maternal obesity on intrapartum outcomes in otherwise low risk women: secondary analysis of the Birthplace national prospective cohort study. BJOG. 2014 Feb;121(3):343-55. doi: 10.1111/1471-0528.12437. Epub 2013 Sep 11. PMID 24034832
- [Result] Silva JC, Amaral AR, Ferreira BD, Petry JF, Silva MR, Krelling PC. [Obesity during pregnancy: gestational complications and birth outcomes.]. Rev Bras Ginecol Obstet. 2014 Nov;36(11):509-513. doi: 10.1590/s0100-720320140005024. Epub 2014 Nov 1. Portuguese. PMID 25493403
- [Result] Zhu T, Tang J, Zhao F, Qu Y, Mu D. Association between maternal obesity and offspring Apgar score or cord pH: a systematic review and meta-analysis. Sci Rep. 2015 Dec 22;5:18386. doi: 10.1038/srep18386. PMID 26692415
- [Result] Bavenas E, Moller C, Bhandarkar P, Mulowooza J, Lofgren J. Predictors of immediate neonatal outcome after cesarean section in Uganda. Int J Gynaecol Obstet. 2022 Jul;158(1):101-109. doi: 10.1002/ijgo.13986. Epub 2021 Nov 8. PMID 34655232